CLINICAL TRIAL: NCT05714618
Title: Magnetic Resonance Imaging Evidence of Cardiac Inflammation Post-Stroke
Brief Title: MR Evidence of Cardiac Inflammation Post-Stroke
Acronym: MIRACLE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: McMaster University (Other); Western University, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: R-21-323
Record Dates: First submitted 2022-01-31; First posted 2023-02-06 (Actual); Last update posted 2024-09-20 (Actual); Status verified 2023-10

CONDITIONS: Stroke, Ischemic; Inflammation; Myocardial Injury
MeSH Terms: conditions — Ischemic Stroke; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases (Ischemic stroke): Left and right middle cerebral artery ischemic stroke: Patients presenting with acute onset focal neurological deficits and DWI-MRI evidence of an acute brain infarct of the left or right middle cerebral artery ischemic stroke.
  Interventions: Diagnostic Test: Gadolinium-enhanced cardiac MRI; Diagnostic Test: B Natriuretic Peptide; Diagnostic Test: Systemic inflammatory markers
- Controls (TIA): Patients with acute focal neurological symptoms without brain infarct on MRI.: Patients presenting with acute onset focal neurological deficits presumed to be of vascular origin, WITHOUT DWI-MRI evidence of an acute brain infarct.
  Interventions: Diagnostic Test: Gadolinium-enhanced cardiac MRI; Diagnostic Test: B Natriuretic Peptide; Diagnostic Test: Systemic inflammatory markers

INTERVENTIONS:
Diagnostic Test: Gadolinium-enhanced cardiac MRI — Cardiac magnetic resonance imaging (MRI) with a protocol designed to measure myocardial inflammation and fibrosis.
Diagnostic Test: B Natriuretic Peptide — Measurement of B Natriuretic Peptide on patients' blood samples at 10 and 60+/-15 days.
Diagnostic Test: Systemic inflammatory markers — Measurement of a panel of 92 systemic inflammatory markers on patients' blood samples at 10 and 60+/-15 days.

SUMMARY:
The present study is an investigator initiated, single-centre, prospective, proof-of-concept cohort study aiming to enroll 44 patients with acute middle cerebral artery (MCA) ischemic stroke, involving the right (n=22) and left (n=22) MCA territories and 24 control patients with acute focal neurological symptoms but no evidence of acute brain infarct on DWI-MRI.

DETAILED DESCRIPTION:
The present study is an investigator-initiated, single-center, prospective cohort study. The study aims to enroll 44 patients with acute/subacute middle cerebral artery (MCA) ischemic stroke. The investigators will compare inflammatory markers among 44 patients with MCA ischemic stroke within 10 days post-stroke vs. 60±15 days post-stroke. Other measures to be determined at both time points include B-Type Natriuretic Peptide and systemic inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

• Acute ischemic stroke in the right or left MCA territory. Acute ischemic stroke is defined as acute onset focal symptoms matching an acute brain infarct documented on Head computed tomography or diffusion-weighted imaging (DWI) MRI of the brain showing restricted diffusion.

Exclusion Criteria:

* History of known atrial fibrillation, prior myocardial infarction, coronary artery disease, heart failure, prior cardiovascular surgery or percutaneous intervention.
* Previous stroke (occurred within 3 months before the index event)
* Impaired renal function defined as a creatinine clearance <97 mL/min in men or <88 mL/min in women, according to the Cockcroft formula.
* hs-TnT >100 on routine acute stroke baseline bloodwork upon admission.
* Clinically or neurologically unstable patients as per the treating physician.
* Ongoing infection or recent infection within the previous 3 months
* Surgery within 3 months before the stroke
* Concurrent and active inflammatory conditions (connective tissue diseases, rheumatological disease, etc.) or use of anti-inflammatory medications
* Pregnancy, Stage IV renal insufficiency, eGFR <30, and any other contraindications to the use of gadolinium.
* Stroke with symptomatic hemorrhagic transformation
* Subjects will be excluded if they fail the LHSC standard MRI screening questionnaire (cardiac pacemakers/wires, aneurysm clips, shunt/surgical clips, shrapnel/bullets, dentures or metal braces, intra-uterine devices, heart valves, ear implants, prostheses, medication patches such as Nicoderm, Habitrol, or Transderm-Nitro, claustrophobia, history of a head or eye injury involving metal fragments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators will include 44 patients with right (n=22) and left (n=22) MCA ischemic stroke. The investigators aim to include at least 50% of female patients. The investigators will include 24 participants in a control group. Participants in the control group will be patients presenting with acute stroke symptoms but no evidence of acute brain infarction on DWI-MRI imaging. Participants will be divided by sex: the investigators aim to enroll 12 female and 12 male participants. The investigators will aim to enroll participants within the same age range as the stroke participants.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2025-06-16 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The severity of left ventricular myocardial inflammation on cardiac MRI within 10 days post-stroke | Within 10 days of stroke onset
  Proportion of left ventricular myocardium showing inflammatory changes on gadolinium-enhanced cardiac MRI
The extent of left ventricular fibrosis measured on gadolinium-enhanced cardiac MRI within 10 days of stroke onset | Within 10 days of stroke onset
  Proportion of left ventricular myocardium showing fibrosis on gadolinium-enhanced cardiac MRI

SECONDARY OUTCOMES:
Changes in left ventricular inflammation measured on gadolinium-enhanced cardiac MRI at 10 and 60±15 days post-stroke | At 60±15 days compared to first 10 days
  Quantification of left ventricular inflammation measured on gadolinium-enhanced cardiac MRI
Change in B-Type Natriuretic Peptide (NT-proBNP) levels in the second measurement performed at 60±15 days post-stroke relative to the plasma sample drawn within 10 days. | At 60±15 days compared to first 10 days
  Change in levels of NT-proBNP between 10 and 60±15 days post-stroke
Change in systemic inflammatory markers between 10 and 60±15 days post-stroke | At 60±15 days compared to first 10 days
  High-performance protein biomarker panel for following 92 inflammatory biomarkers in pg/mL
  ADA; ARTN; AXIN1; NGF; CCL13; CCL19; CCL2; CCL20; CCL23; CCL25; CCL28; CCL3; CCL4; CCL7; CCL8; CXCL10; CXCL11; CXCL5; CXCL6; CXCL9; CDCP1; CASP8; CST5; DNER; CCL11; EIF4EBP1; FGF19; FGF21; FGF23; FGF5; FLT3LG; CX3CL1; GDNF; CXCL1; HGF; IFNG; IL1A; IL10; IL10RA; IL10RB; IL12B; IL13; IL15RA; IL17A; IL17C; IL18; IL18R1; IL2; IL2RB; IL20; IL20RA; IL22RA1; IL24; IL33; IL4; IL5; IL6; IL7; CXCL8; MMP1; KITLG; LIF; LIFR; LTA; CSF1; SIRT2; CD244;NTF3;NRTN;OSM;CD274;S100A12;TGFA;STAMBP;SLAMF1;MMP10;SULT1A1;CD6;CD5;CD8A;TSLP;TGFB1;TNF;TNFSF10;TNFSF11;TNFSF12;TNFSF14;TNFRSF11B;CD40;TNFRSF9;PLAU;VEGFA
Changes in left atrial inflammation measured on gadolinium-enhanced cardiac MRI at 10 and 60±15 days post-stroke | At 60±15 days compared to first 10 days
  Quantification of left atrial inflammation measured on gadolinium-enhanced cardiac MRI
Changes in left atrial fibrosis measured on gadolinium-enhanced cardiac MRI at 10 and 60±15 days post-stroke | At 60±15 days compared to first 10 days
  Quantification of left atrial fibrosis measured on gadolinium-enhanced cardiac MRI

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Sposato, MD, Principal Investigator — London Health Sciences Center, Western University
Locations (1):
- Heart & Brain Lab, Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided